CLINICAL TRIAL: NCT05652790
Title: Pragmatic Prospective, Multicentre Feasibility Non-randomised Controlled Trial on Enhanced Rehabilitation for Poly & Lower Extremity Trauma (PROPERLY Trial)
Brief Title: Enhanced Rehabilitation After Major Trauma (PROPERLY)
Acronym: PROPERLY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: Northern Care Alliance NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B01762
Record Dates: First submitted 2022-11-25; First posted 2022-12-15 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Major Trauma
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Pragmatic Prospective, multicentre feasibility non-randomised controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Rehabilitation Programme (ERP) (Experimental): 60-120 MINUTES OF ENHANCED REHABILITATION
  Manual Therapy Hydrotherapy Exercise Strength and Conditioning Programmes Gait re-education Pilates/ Yoga Cognitive and Vocational Rehabilitation Occupation Therapy Interventions eg. Anxiety Management, Pacing, Cognitive Behavioural Therapy
  Interventions: Procedure: Enhanced Rehabilitation Programme
- Standard Care (Other): Standard care received at usual NHS facility
  Interventions: Procedure: Standard Care

INTERVENTIONS:
Procedure: Enhanced Rehabilitation Programme — The ERP would be offered at least two sessions, each lasting 60-120 minutes per week, delivered in the Manchester Institute of Health and Performance. Interventions may include a combination of the following depending on the individual patient needs.
  Manual Therapy Hydrotherapy Exercise Strength and Conditioning Programmes Gait re-education Pilates/ Yoga Cognitive and Vocational Rehabilitation Occupation Therapy Interventions eg. Anxiety Management, Pacing, Cognitive Behavioural Therapy
  Other Names: ERP
  Arms: Enhanced Rehabilitation Programme (ERP)
Procedure: Standard Care — Standard care received at usual NHS facility
  Other Names: SC
  Arms: Standard Care

SUMMARY:
The goal of this study is to assess the feasibility of recruitment, and barriers to delivery of an enhanced rehabilitation service, in patients surviving major trauma.

The main questions it aims to answer are:

are the investigators able to recruit patients to a research study are the investigators able to retain patients in the research study are the investigators able to identify appropriate primary outcome measures are the investigators able to identify barriers to future large-scale definitive trial or service delivery Participants will would be offered at least two sessions of the Enhanced Rehabilitation Programme (ERP), each lasting 60-120 minutes per week, delivered in the Manchester Institute of Health and Performance (MIHP).

Participants not willing to travel to the MIHP, or declining to engage in the ERP, will be asked to join the Standard Care (SC) group. This group will provide questionnaire data and clinical outcome measure collection with their usual place of therapy.

Researchers will compare the ERP group and the SC groups to assess any additional benefits to the ERP.

DETAILED DESCRIPTION:
The investigators will aim to recruit 25 participants for the ERP and 25 participants in SC (50 in total) who will go through a series of quantitative functional assessments and patient reported outcome measures, at baseline (at the beginning of the programme), middle (3 months), on discharge from the programme (usually 6 months). If patients are discharged earlier, assessments will be performed at the discharge visit.

Assessments using PROMS will be conducted at baseline (at the beginning of the programme), middle (3 months), on discharge from the programme (usually 6 months), and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants over 18 years old
* Registered GP in Greater Manchester or Greater Manchester Resident.
* Polytrauma or one or more complex /severe isolated injury
* Rehabilitation goals (e.g., mobility, function, job retention/ return to work) identified using shared decision-making process
* Patient able to enter programme 6-30 months post injury.
* For the ERP patients willing to travel to the MIHP for their evaluation and treatment twice a week.
* Participants with lower limb injuries that continue to have functional impairment.
* Participants deemed well and safe enough to participate by clinical teams.
* Normal ECG if previously reported to have abnormal ECG
* Participants willing to consent to follow up over 12 months
* Participants with the capacity to consent to the study.
* Fully healed wounds and bone healed sufficiently to allow at least partial weight bearing

Exclusion Criteria:

* Participants under the age of 18
* Participants unable to provide informed consent
* Participants with multiple pre-existing comorbidities that affect ability to participate in enhanced rehabilitation such as cognitive impairment, unstable angina.
* Central motor neurological impairment affecting ability to participate in an enhanced rehab programme
* Absence of functional disability affecting gait and / or function.
* Plans for further surgery that will impact on gait or function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Recruitment & retention into both arms of the trial | 12 months
  Number of patients recruited to ERP

SECONDARY OUTCOMES:
EQ-5D-L | baseline, 3, 6 months and 12 months.
  Functional impairment outcome measure
  The lowest score of 0 indicates no functional impairment and a score of 4 indicates significant impairment. The category responses are not combined.
  Using a continuous scale on a 20cm vertical visual analogue scale (VAS) a score of 100 means 'the best health imaginable and a score of 0 means 'the worst health imaginable.' EQ5DL Scores at different timepoints are compared to show changes in health over time.
PHQ9 | baseline, 3, 6 months and 12 months
  Patient Health Questionnaire 9 The Patient Health Questionnaire-9 (PHQ-9) is a brief psychological screening instrument designed to measure symptoms of depression in healthcare settings.
  It contains 9 questions that help identify patients with clinically meaningful symptoms of depression. Patient responses are scored 0-3 with 0 representing "not at all" and 3 indicating "nearly every day;" thus, the PHQ-9 contains a total score range of 0-27
GAD7 | baseline, 3, 6 months and 12 months
  General Anxiety and Depression Score 7 is a self-administered patient questionnaire used as a screening tool and severity measure for generalised anxiety disorder (GAD).
  The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions.
  Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater.
LEFS | baseline, 3, 6 months and 12 months
  Lower Extremity Functional Scale (LEFS) determines functional status in patients suffering from lower extremity disorders and disabilities.
  This health tool evaluates the ability of the subject to perform daily activities. It comprises of a list of 20 everyday tasks and is used by clinicians as a measure of functional status and in setting goals and monitoring progress in different conditions. Participants rate the level of difficulty as follows
  * Extreme difficulty or unable to perform activity (0 points);
  * Quite a bit of difficulty (1 point);
  * Moderate difficulty (2 points);
  * A little bit of difficulty (3 points);
  * No difficulty (4 points);
  The maximum score obtainable is 80 points which signifies complete function and the lowest score is 0 which indicates very low function. All LEFS scores are then awarded as number of points out of the total of 80.
Two-minute walk test | baseline, 3, 6 months and 12 months
  the Two-minute walk test is a simple functional test that evaluates submaximal exercise, test used to assess aerobic capacity and endurance. The distance covered over a time of 2 minutes is used as the outcome by which to compare changes in performance capacity
30SSTS | baseline, 3, 6 months and 12 months
  30 Second sit to stand test
  30 Second Sit to Stand Test (also known as 30 second chair stand test - 30CST), is for testing leg strength and endurance (Rikli & Jones 1999), where patients are asked to repeat sitting and standing as quickly as possible without the aid of their arms on a standardised seat. The total number of completed Sit to Stands is recorded as the measure.
Y Balance test | baseline, 3, 6 months and 12 months
  The Lower Quarter Y Balance Test (LQYBT) is a tool used to test a person's risk for injury by evaluating balance, gait stability and strength.
  Patients stand on one leg while reaching out in 3 different directions with the other lower extremity, the 3 reaches yield a "composite reach distance" or composite score used to predict injury.
Pain score | baseline, 3, 6 months and 12 months
  A Numerical Pain Rating Scale (NRS) will be used to assess patients pain throughout the programme. (0-100)
  - 0 is worse pain 100 is no pain (Jensen et al, 1995)
ABCS | baseline, 3, 6 months and 12 months
  Activities Specific Balance Confidence Scale is a structured questionnaire that measures an individual's confidence during ambulatory activities without falling or experiencing a sense of unsteadiness.
  The ABCS is a 16-item questionnaire where patients' rate their confidence while doing activities.
  Scoring from 0-100 (0 is no confidence and 100 is full confidence)
  Lower than 50 %: low level of physical functioning 50-80 %: moderate level of physical functioning Above 80 %: high level of physical functioning
Participant and Practitioner experience | Baseline and 6 months
  Participant and Practitioner interviews to evaluate
  * Participants with multiple pre-existing comorbidities that affect ability to participate in enhanced rehabilitation such as cognitive impairment, unstable angina, foot ulcers, inflammatory arthritis, injury
  * Central neurological impairment
  * Absence of functional disability affecting gait.
  * Awaiting further surgery that will affect function

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wong, MD, Study Chair — National Health Service, United Kingdom
Locations (1):
- Manchester University NHS Foundation Trust - St Mary's, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
no plan